CLINICAL TRIAL: NCT01250067
Title: Motor-related Cortical Potential in Patients With Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NSC92-2314-B-039-016
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2005-09

CONDITIONS: Essential Tremor; Movement-related Cortical Potentials
MeSH Terms: conditions — Essential Tremor

INTERVENTIONS:
Procedure: Motor-related cortical potential (Procedure)

SUMMARY:
In this proposal, in addition to the conventional MRCP recording, the dipoles and sources of the different subcomponents of MRCP will also be analyzed with the brain electric source analysis (BESA) to evaluate the difference in the solutions and source strength underlying the MRCP between normal controls and patients with ET.

DETAILED DESCRIPTION:
Essential tremor (ET) is a common disorder with unknown etiology and pathogenesis. Typically described as a postural tremor, ET often has a marked kinetic component suggesting cerebellar involvement in the pathogenesis of the tremor. The assumption has been illustrated by both positron emission tomography and functional magnetic resonance imaging studies, which revealed that blood flow and activity of the cerebellum were increased in ET patients as compared to the normal controls. In contrast to the cumulative body of imaging evidence, the physiological bases to link the ET and cerebellar functional alternation are scarce. Studies with tandem gait analysis have revealed 25% abnormality of ET patients and surface electromyographic study has found a delay in the second agonist burst during rapid wrist movements suggesting the possible role of cerebellar functional alternation in the generation of ET. In addition, since the tremor of ET tends to appear in the movement ignition or during postural maintenance, it is conceivable that this sort of tremor might exert certain impact on the programming and preparation of the limb movement. Thus it would be appropriate to adopt a tool, which can concomitantly assess the cerebellar function and movement preparation, to investigate the patients with ET. In this proposal, we will record movement-related cortical potentials (MRCP) in ET patients. MRCP is a slow negative shift starting 1-1.5 sec before volitional movement. It consists of at least 3 subcomponents, the Bereitschaftspotential, the negative slope, and the motor potential. The generators crucial for the generation of MRCP include cerebellum, motor and motor association cortex. Thus MRCP seems to be an appropriate tool to assess the patients with ET, in whom the trivial cerebellar functional alternation could be responsible for the tremor generation and motor preparation might be hampered concomitantly. In this proposal, in addition to the conventional MRCP recording, the dipoles and sources of the different subcomponents of MRCP will also be analyzed with the brain electric source analysis (BESA) to evaluate the difference in the solutions and source strength underlying the MRCP between normal controls and patients with ET.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral postural tremor with or without kinetic tremor involving hands or forearms, which is visible and persistent, and long-standing in duration (>5 years). Tremor involving body parts other than upper limbs may be present, the tremor may be asymmetrical, amplitude may fluctuate, and the tremor may or may not produce disability.

Exclusion Criteria:

* Neurological signs, except for Froment's sign
* Causes of enhanced physiologic tremor
* Concurrent or recent exposure to tremorgenic drugs
* Direct or indirect trauma to the central and peripheral nervous system
* Historical or clinical evidence of psychogenic origins of tremor
* Convincing evidence of sudden onset or evidence of stepwise deterioration

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Chon-Haw Tsai, MD, Ph.D., Principal Investigator — Department of Neurology, China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan